CLINICAL TRIAL: NCT02066688
Title: A Randomize Controlled Trial of Folic Acid, Calcium and Vitamin D in Preventing Colorectal Polyps and Colorectal Cancer
Brief Title: Study of Folic Acid, Calcium and Vitamin D in Preventing Colorectal Polyps and Colorectal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Director of Department of Gastroenterology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SQ2011SF12RJ; SQ2011SF12-20121010 (Registry Identifier: Ying-xuan Chen)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folic Acid; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FA (Experimental): Patients receive oral folic acid pill 1 mg daily for 36 months in the absence of unacceptable toxicity or any other adverse effects (FA Arm).
  Interventions: Drug: folic acid
- FA+Ca (Experimental): Patients receive oral folic acid pill 1 mg+ calcium 1200mg +vitamin D3 250 IU daily for 36 months in the absence of unacceptable toxicity or any other adverse effects(FA+Ca arm).
  Interventions: Drug: folic acid calcium vitamin D3
- Ca (Experimental): Patients receive oral calcium 1200mg +vitamin D3 250 IU daily for 36 months in the absence of unacceptable toxicity or any other adverse effects (Ca Arm).
  Interventions: Drug: calcium
- blank control group (Placebo Comparator): Patients receive oral placebo once daily for 36 months in the absence of unacceptable toxicity or any other adverse effects.

INTERVENTIONS:
Drug: folic acid — Patients receive oral folic acid 1mg daily for 36 months in the absence of unacceptable toxicity or any other adverse effects.
  Arms: FA
Drug: folic acid calcium vitamin D3 — Patients receive oral folic acid 1mg + calcium 1200mg +vitamin D3 250 IU daily for 36 months in the absence of unacceptable toxicity or any other adverse effects .
  Arms: FA+Ca
Drug: calcium — calcium 1200mg/d + vitamin D3 250 IU/d daily supplements
  Arms: Ca

SUMMARY:
Folic acid (FA) and its derivatives (folate) which play a role in nucleotide synthesis and methylation reactions as well as calcium and vitamin D are assumed to be effective in the prevention of colorectal polyps and Colorectal cancer (CRC). The aim of this study is to investigate the roles of FA as well as calcium and vitamin D in the prevention of CRC.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) affects approximately one million people each year with a five-year survival rate of 62% . Considerable interest has recently been focused on the relationship between the chemoprevention of colorectal polyps/CRA and CRC. Therefore, the use of nutritional compounds which are usually less afflicted with the risk of severe side effects for colorectal adenoma (CRA) prevention and health maintenance is an emerging field.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 50-80 years
* Patients had undergone complete colonoscopy with no adenoma found
* Those who voluntarily sign the consent form after being fully informed and understanding the purpose and procedures of the study, characters of the disease, effect of medications, methods of related examinations, and potential risk/benefits of the study

Exclusion Criteria:

* Patients who are hypersensitive or intolerant to the drugs
* Patients who are intolerant to another colonoscopy examination
* Pregnant women, woman during breast-feeding period, or women with expect pregnancy
* Patients with diabetes mellitus, severe heart or renal disease，or cancer history
* Patients with malignant neoplasm, or suspicious colorectal cancer
* Patients who are not able to cooperate
* Individuals who are involved in designing, planning or performing this experiment
* Patients with medical conditions who are not appropriate to participate the study
* Patients who are take aspirin or cyclooxygenase 2 inhibitor （COX2）.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate the incidence of colorectal adenoma (CRA) after Folic acid, calcium and vitamin D intervention. | baseline and 3 years

SECONDARY OUTCOMES:
the incidence of advanced colorectal adenoma (A-CRA) after Folic acid, calcium and vitamin D intervention. | baseline and 3 years
changes in serum calcium | baseline and 3 years
changes in serum FA | baseline and 3 years
the incidence of colorectal cancer (CRC) after Folic acid, calcium and vitamin D intervention. | baseline and 3 years
changes in clinical symptoms scores (positive immunochemical fecal occult blood test (iFOBT), diarrhea, or constipation et al) | baseline and 3 years
differences in Histological types of CRA OR CRC | baseline and 3 years

OTHER OUTCOMES:
Changes in routine blood count, urine and stool routine test, liver and kidney functions | baseline and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jing-yuan Fang, MD., Ph D., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Renji Hospital, Shanghai, China